CLINICAL TRIAL: NCT00452608
Title: Use of Statins in Modulation of Inflammatory Answer in Septic Patients
Brief Title: Statin for Immunomudulation in Sepsis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Nadine Clausell, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05589
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2009-06-26 (Estimated); Status verified 2009-06

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- amido pill (Placebo Comparator)
  Interventions: Drug: amido pill
- atorvastatina (Experimental): atrovastatina 80 mg/d by mouth for 10 days
  Interventions: Drug: atorvastatina

INTERVENTIONS:
Drug: amido pill — one pill of amido/d by mouth for 10 days
  Arms: amido pill
Drug: atorvastatina — atorvastatina 80 mg/day by mouth for 10 days
  Arms: atorvastatina

SUMMARY:
The purpose of this study is to determine whether atorvastatin can improve the inflammatory answer in the septic patients

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of several sepsis or shock septic
* no more than twenty four hours than diagnosis

Exclusion Criteria:

* use of statins in the last thirty days
* unequivocal indication for statin treatment
* active treatment with imunosuppressors drugs
* High risk of rhabdomyolysis: multiple trauma, crush injuries, baseline creatinine kinase > three times upper limit of normal
* diagnosis of AIDS
* unable to receive enteral medications
* pregnancy
* expected survival of less than 48 hours

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-12; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
action in inflammmatory biologic makers | 24h; 72h; 10 days
valuation of flow-mediated vasodilation of the brachial artery | 24h; 72; 10 days

SECONDARY OUTCOMES:
mortality | at end
time of permanence in intensive care unity | at end
time of permanence in mechanical ventilation | at end

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Clausell, Principal Investigator — Federal University of Rio Grande do Sul - Brazil
Locations (1):
- HCPA - Clinical Hospital fo Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil